CLINICAL TRIAL: NCT00072826
Title: Atorvastatin Therapy To Improve Endothelial Function in Sickle Cell Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040032; 04-CC-0032
Record Dates: First submitted 2003-11-10; First posted 2003-11-11 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2015-12-07

CONDITIONS: Sickle Cell Disease
Keywords: 3-hydroxy-3-methlglutaryl (HMG); Inhibitors; Endothelial Function; Leukocyte Gene Expression; Statins; Atorvastatin; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Oxypurinol; omega-N-Methylarginine; Acetylcholine

INTERVENTIONS:
Drug: Oxypurinol
Drug: L-NMMA
Drug: Acetylcholine

SUMMARY:
This study will examine the effects of oral atorvastatin on the linings of blood vessels in patients with sickle cell disease, plus the agent's effect on blood markers of inflammation and blood vessel function. Sickle cell disease is a recessive genetic disorder and the most common genetic disease affecting African Americans. Inherited are abnormal genes that make hemoglobin, the substance within red blood cells that carries oxygen from the lungs to the body. In the disease, sickle hemoglobin leads to rigidity or hardness of the red cells, causing obstruction in small blood vessels, inflammation, and injury to organs when the flow of blood to them is blocked. Some medications already prescribed for other diseases, such as atorvastatin, which is used for lowering cholesterol levels, can improve blood flow.

Patients 18 to 65 years of age who have sickle cell disease, who have not had an acute pain episode within the previous week, and who are not pregnant or lactating may be eligible for this study. They will undergo a complete medical history; physical examination; baseline blood tests; and echocardiogram, in which an ultrasound wand is placed against the chest wall to get images inside the heart and blood vessels.

In addition, patients will have blood flow studies. During the procedure, they will lie in an adjustable reclining chair for 5 to 6 hours. There will be 20- to 30-minute rests between specific activities and blood samples will be drawn intermittently for testing. Small tubes will be placed in the artery of the forearm at the inside of the elbow. Normal saline will be infused into one tube. A small pressure cuff will be applied to the wrist and a larger cuff to the upper arm. Both cuffs will be attached to an inflation device. A device like a rubber band, a strain gauge, will be placed around the widest part of the forearm. When the pressure cuffs are inflated, blood will flow into the arm, stretching the gauge proportion to blood flow, and information will be recorded. Then light reflected from the patients' hand and the blood flow in the forearm will be measured. Activity of the genes in the white blood cells will be measured as well. Small amounts of sodium nitroprusside, widely used to reduce blood pressure in people with dangerously high blood pressure, will be injected and blood flow will be measured. Later, small amounts of acetylcholine will be injected. It usually causes blood vessels to expand. After that, small amounts of L-NMMA will be injected. It usually decreases local blood flow by blocking the production of nitric oxide in the cells lining the arm's blood vessels. Then acetylcholine combined with L-NMMA will be injected. After that, oxypurinol, an agent taken by many patients to prevent gout, will be injected. The procedures will be repeated, with oxypurinol given along with each of the agents, and the measurement of blood flow in the forearm will be measured after each drug combination.

Afterward, patients will be treated for 4 weeks at home with oral atorvastatin. They will be asked to visit the Clinical Center every 2 weeks for collection of blood samples and an examination. After 4 weeks of taking atorvastatin orally, they will be asked to return to repeat the blood flow studies, but only the first half will be conducted. The part using oxypurinol will not be needed. Regarding some of the blood samples collected during the study, there will be an examination of the genes found in the white blood cells. Specific attention will go to those genes that make proteins for cell-to-cell interaction and inflammation, plus those that cause blood cells to stick to the lining of blood vessels.

DETAILED DESCRIPTION:
Sickle cell disease is an autosomal recessive disorder and the most common genetic disease affecting African-Americans. Approximately 0.15% of African-Americans are homozygous for sickle cell disease, and 8% have sickle cell trait. Hemoglobin S polymerization leads to red cell rigidity, microvascular obstruction, inflammation, and end-organ ischemic injury. Our published data indicate that up to 50% of sickle cell patients have endothelial dysfunction due to impaired bioavailability of endogenous nitric oxide. Our studies indicate that this is due in large part to scavenging of nitric oxide by cell-free hemoglobin, with additional nitric oxide inactivation by superoxide. This suggests that therapies directed at restoring NO bioavailability might be beneficial. In patients with atherosclerotic vascular disease, the statin family of 3-hydroxy-3-methylglutaryl (HMG) CoA reductase inhibitors significantly reduce stroke and myocardial infarction and restore endothelial-dependent relaxation of conducting arteries. Furthermore, statin therapy has now been clearly shown to reduce C-reactive protein levels and clinical events in patients with coronary artery disease independent of the effects on lipoproteins. The ability of statins to correct vascular inflammation and endothelial dysfunction makes this class of agents attractive to attempt to reverse these features of sickle cell pathobiology. This trial will aim to 1) establish the effects of oral atorvastatin treatment on endothelial-dependent relaxation in patients with sickle cell disease and endothelial dysfunction; 2) establish the effect of therapy on peripheral blood markers of inflammation and vascular function, and peripheral blood proteome and transcriptome profiles; and 3) investigate whether superoxide produced through xanthine oxidase limits nitric oxide bioavailability in patients with sickle cell disease.

In order to control for the possibility that advancing age, gender and ethnicity may influence vascular reactivity, we will also enroll age and gender-matched African-American controls in the baseline forearm blood flow portion of this study.

ELIGIBILITY:
* ELIGIBILITY:

All volunteer subjects must be at least 18 years of age and have provided informed, written consent for participation in this study. Eligibility in the study is determined prior to enrollment on the basis of the following inclusion and exclusion criteria.

INCLUSION CRITERIA FOR CONTROLS:

For each enrolled study patient with sickle cell disease, we will recruit an African-American healthy control subject of the same gender, within 3 years of age older or younger than the matched patient.

INCLUSION CRITERIA FOR SICKLE CELL COHORT:

Males or females 18 to 65 years of age.

Diagnosis of sickle cell disease (electrophoretic or HPLC documentation of hemoglobin S only phenotype is required).

Hemoglobin must be 6-9 g/dL with an absolute reticulocyte count greater than 95,000/microL, or hemoglobin greater than 9 g/dL with no requirement for reticulocyte count.

Plasma soluble VCAM level above median value for sickle cell patients defined by assays performed in our laboratory on the blood of sickle cell patients seen in our program or tricuspid regurgitant jet velocity (determined by Doppler echocardiography) greater than 2.4 m/sec or has had a subnormal response to L-NMMA or sodium nitroprusside infusion on a previous forearm blood flow study.

EXCLUSION CRITERIA FOR SICKLE CELL COHORT:

Clinically unstable sickle cell disease defined as having an acute pain crisis within the last week.

Current pregnancy or lactation.

Conditions that may independently affect endothelial function:

Diabetes mellitus or fasting blood sugar greater than 120 mg/dL

Cigarette smoking within one month

Hypertension (diastolic blood pressure greater than 90 mmHg)

Serum creatinine greater than 1.5 mg/dL

Serum alanine aminotransferase (ALT) greater than 3 times the upper limit of normal. (AST elevation will not be used as an exclusion criteria, since this is elevated in normal sickle cell patients due to red cell lysis, even without liver injury)

Hemoglobin less than or equal to 6 g/dL; however, patients may return for evaluation at a later date.

Recent transfusion (last 4 weeks).

No aspirin or non-steroidal anti-inflammatory drugs (NSAIDs) for one week and no caffeine the day of the study. Patients on opiates or acetaminophen will not be excluded.

Subjects taking sildenafil, vardenafil, L-arginine, fibrates (e.g., clofibrate, gemfibrozil, or fenofribrate) or inhaled nitric oxide within the last week will be excluded from the study.

Subjects taking any statin drug (e.g., fluvastatin, lovastatin, pravastatin, or simvastatin) within the last four weeks will be excluded from the study.

Subjects taking drugs with known clinically significant metabolic interactions with statins (via metabolism through cytochrome P450 3A4):

Ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, azithromycin, cyclosporine, tacrolimus, fibric acid derivatives, niacin (nicotinic acid).

Subjects who have obstructive or vasospastic vascular disease.

Subjects with significant cardiac disease and/or ECG abnormalities.

Subjects with significant hypotension.

Women who do not use two forms of birth control while participating in this study.

EXCLUSION CRITERIA FOR CONTROLS:

Current pregnancy or lactation.

Conditions that may independently affect endothelial function:

* Diabetes mellitus or fasting blood sugar greater than 120 mg/dL
* Cigarette smoking within one month
* Hypertension (diastolic blood pressure greater than 90 mmHg)

Serum creatinine greater than 1.5 mg/dL

Serum alanine aminotransferase (ALT) greater than 3 times the upper limit of normal.

Hemoglobin less than 12 g/dL; however, patients may return for evaluation at a later date.

No aspirin or non-steroidal anti-inflammatory drugs (NSAIDs) for one week and no caffeine the day of the study. Patients on opiates or acetaminophen will not be excluded.

Subjects taking sildenafil, vardenafil, L-arginine, fibrates (e.g., clofibrate, gemfibrozil, or fenofribrate) or inhaled nitric oxide within the last week will be excluded from the study.

Subjects taking any statin drug (e.g., fluvastatin, lovastatin, pravastatin, or simvastatin) within the last four weeks will be excluded from the study.

Subjects who have obstructive or vasospastic vascular disease.

Subjects with significant cardiac disease and/or ECG abnormalities.

Subjects with significant hypotension.

Subjects with any known form of hemolytic anemia, including sickle cell disease (Hb SS, SC, S-beta-thalassemia, or other known sickling syndromes; sickle trait will NOT be excluded).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2003-11-04; Primary Completion 2007-08-24 (Actual); Study Completion 2007-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F Tisdale, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Quyyumi AA, Dakak N, Andrews NP, Husain S, Arora S, Gilligan DM, Panza JA, Cannon RO 3rd. Nitric oxide activity in the human coronary circulation. Impact of risk factors for coronary atherosclerosis. J Clin Invest. 1995 Apr;95(4):1747-55. doi: 10.1172/JCI117852. PMID 7706483
- [Background] Panza JA, Casino PR, Kilcoyne CM, Quyyumi AA. Role of endothelium-derived nitric oxide in the abnormal endothelium-dependent vascular relaxation of patients with essential hypertension. Circulation. 1993 May;87(5):1468-74. doi: 10.1161/01.cir.87.5.1468. PMID 8491001
- [Background] Britten MB, Zeiher AM, Schachinger V. Clinical importance of coronary endothelial vasodilator dysfunction and therapeutic options. J Intern Med. 1999 Apr;245(4):315-27. doi: 10.1046/j.1365-2796.1999.00449.x. PMID 10356593